CLINICAL TRIAL: NCT00248547
Title: A Pilot Study of Aprepitant vs. Placebo Combined With Standard Antiemetics for the Control of Nausea and Vomiting During Hematopoietic Cell Transplatation(HCT)
Brief Title: Aprepitant in Preventing Nausea and Vomiting in Patients Who Are Undergoing a Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Joseph Bubalo, PharmD, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CDR0000445452; OHSU-HEM-03074-L (Other: OHSU Knight Cancer Institute); OHSU-1057 (Other: OHSU IRB); MERCK-OHSU-HEM-03074-L (Other: Merck)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: nausea and vomiting; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent small lymphocytic lymphoma; recurrent malignant testicular germ cell tumor; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage II ovarian epithelial cancer; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III ovarian epithelial cancer; stage III small lymphocytic lymphoma; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV ovarian epithelial cancer; stage IV small lymphocytic lymphoma; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Neuroblastoma; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Testicular Neoplasms; Leukemia, Hairy Cell; Multiple Myeloma; Breast Neoplasms | interventions — Aprepitant; Dexamethasone; Calcium Dobesilate; Ondansetron; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant (Active Comparator)
  Interventions: Drug: aprepitant; Drug: dexamethasone; Drug: ondansetron
- sugar pill (Placebo Comparator): Loading dose of 125 mg capsule once a day for one day, then maintenance dose of 80 mg capsule daily through Day +4 of Bone Marrow Transplant
  Interventions: Drug: dexamethasone; Drug: ondansetron; Drug: placebo

INTERVENTIONS:
Drug: aprepitant — Loading dose of 125 mg capsule once a day for one day, then maintenance dose of 80 mg capsule daily through Day +4 of Bone Marrow Transplant
  Other Names: Emend
  Arms: Aprepitant
Drug: dexamethasone — For Cyclophosphamide Total Body Irradiation(CyTBI) patients: Dexamethasone study drug 1 capsule PO daily, 1 hour prior to chemotherapy with aprepitant on total body irradiation(TBI) and cyclophosphamide chemotherapy days; For Busulfan Cyclophosphamide(BuCy) patients: Dexamethasone 1 capsule orally once daily, discontinue after last dose of chemotherapy.
  Other Names: Decadron
Drug: ondansetron — For CyTBI patients: Ondansetron 8 mg orally evert 12 hours, begin 1 hour prior to first TBI dose and discontinue after last dose; then Ondansetron 8 mg IV every 12 hours X 4 doses, begin 30 minutes prior to first cyclophosphamide chemotherapy; For BuCy patients: Ondansetron 8 mg orally every 6 hours, begin 1 hour prior to first busulfan dose and discontinue after last busulfan dose is given. then: Ondansetron 8 mg IV Q 12 hours X 4 doses, begin 30 minutes prior to first cyclophosphamide chemotherapy
  Other Names: Zofran
Drug: placebo — Loading dose of 125 mg capsule once a day for one day, then maintenance dose of 80 mg capsule daily through Day +4 of Bone Marrow Transplant
  Other Names: placebo, sugar pill
  Arms: sugar pill

SUMMARY:
RATIONALE: Antiemetic drugs, such as aprepitant, ondansetron, and dexamethasone, may help lessen or prevent nausea and vomiting in patients undergoing a stem cell transplant.

PURPOSE: This randomized clinical trial is studying aprepitant, ondansetron, and dexamethasone to see how well they work compared to placebo, ondansetron, and dexamethasone in preventing nausea and vomiting in patients who are undergoing a stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of standard antiemetic therapy comprising ondansetron and dexamethasone combined with either aprepitant or placebo in controlling nausea and vomiting, as determined by the number of retch/emesis-free days, in patients undergoing hematopoietic stem cell transplantation.

Secondary

* Determine the safety of aprepitant in these patients.
* Compare nausea, appetite, taste changes, nutritional intake, and mucositis in patients treated with these regimens.
* Determine the pharmacokinetics of cyclophosphamide, carboxyethylphosphoramide mustard, hydroxycyclophylamide, and aprepitant in these patients.

OUTLINE: This is a randomized, placebo-controlled, single-blind, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning on the first day of conditioning chemotherapy, patients receive oral aprepitant once daily and standard antiemetic therapy comprising oral or IV ondansetron and oral dexamethasone.
* Arm II: Patients receive oral placebo once daily and standard antiemetic therapy as in arm I.

In both arms, treatment continues until day 4 after stem cell transplant in the absence of unacceptable toxicity.

After completion of study therapy, patients are followed until day 18.

PROJECTED ACCRUAL: A total of 40 patients (20 per treatment arm) will be accrued for this study.

ELIGIBILITY:
Inclusion:

* 18 years of age or greater
* must be scheduled for an autologous or allogeneic bone marrow or peripheral stem cell transplant
* Eastern Cooperative Oncology Group(ECOG) performance status < or = 2
* patients must have signed informed consent
* must be able to swallow tablets and capsules
* must be receiving a cyclophosphamide containing regimen.

Exclusion:

* patient has known sensitivity to aprepitant, ondansetron, or dexamethasone
* patient has received another investigational drug in the past 30 days
* patient has had emesis or requires antiemetic agents in the 48 hours prior to beginning conditioning therapy
* patient has taken neurokinin-1 antagonists for 14 days prior to enrollment
* patient is pregnant, has a positive serum human chorionic gonadotropin(hCg) or is lactating
* patient has serum creatinine level > or = 2*ULN
* patient has severe hepatic insufficiency (Child-Pugh score >9)
* patient drinks > 5 drinks/day for the last year
* patient with concurrent illness requiring systemic corticosteroid use other than planned dexamethasone during conditioning therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Bubalo, PharmD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inpatients receiving allogeneic bone marrow transplants who were to get either Busulfan/Cytoxan or Cytoxan/Total Body Radiation as conditioning regimen.
Period: Overall Study
Arm/Group | Aprepitant | Placebo
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12.9) | 46 (13) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Emesis Free Participants During the Study Period.
Description: To compare the efficacy of aprepitant plus standard therapy to placebo plus standard therapy in control of nausea and vomiting during conditioning therapy for autologous or allogeneic hematopoietic stem cell transplantation (HSCT) as defined by the number of retch/emesis free days during the study period
Time Frame: Up to three weeks
Measure: Number; unit: Participants
Groups:
- Placebo (Sugar Pill): Loading dose of 125 mg capsule once a day for one day, then maintenance dose of 80 mg capsule daily through Day +4 of Bone Marrow Transplant
Arm/Group | Aprepitant | Placebo (Sugar Pill)
Number analyzed (Participants) | 20 | 20
Participants | 13 | 5
Statistical Analysis 1: Comparison: Aprepitant vs Placebo (Sugar Pill); Test type: Superiority or Other; p = 0.041, Wilcoxon Rank Sum Test

2. Secondary Outcome: Safety in Transplant Population
Description: To assess the safety of aprepitant in the bone marrow transplant population
Time Frame: Up to three weeks
Reporting Status: Not Posted

3. Secondary Outcome: Effects on Nausea, Appetite and Taste Changes
Description: To assess the effects of aprepitant on nausea, appetite, and taste changes, (via visual analogue scale [VAS]), nutritional intake, and mucositis in the bone marrow transplant population.
Time Frame: Up to three weeks
Reporting Status: Not Posted

4. Secondary Outcome: Pharmacokinetic Interaction
Description: To assess the potential for aprepitant and cyclophosphamide to interact pharmacokinetically in a significant manner to change blood levels of aprepitant, cyclophosphamide, hydroxycyclophosphamide or CEPM.
Time Frame: Up to three weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Aprepitant | Placebo
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant (N=20) | Placebo (N=20)
Subileus (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No